CLINICAL TRIAL: NCT00646724
Title: Cotransplantation of Islet and Mesenchymal Stem Cell in Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: FUZHOU GENERAL HOSPITAL, FUZHOU GENERAL HOSPITAL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fuzhough0712; fuzhough0712
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islets of Langerhans Transplantation; Mesenchymal Stem Cells; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): cotransplantation of islet and mesenchymal stem cell
  Interventions: Biological: cotransplantation of islet and mesenchymal stem cell

INTERVENTIONS:
Biological: cotransplantation of islet and mesenchymal stem cell — islet of allograft and MSCs of autograft

SUMMARY:
The study evaluates the safety and efficacy of Cotransplantation of Islet and Mesenchymal Stem Cell in Type 1 Diabetic Patients. The researchers hypothesize that additional Mesenchymal Stem Cell infusion can benefit the promising clinical islet transplantation through the following mechanisms: protection of islet from inflammatory damage, immunological modulation, engraftment promotion, thus decrease or eliminate the need of exogenous insulin and improve β-cell function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 60 years of age
* Ability to provide written informed consent
* Manifest signs and symptoms that are severe enough to be incapacitating
* Patients with poor diabetes control (HbA1c > 7% but < 12%)
* Progressive diabetic complications

Exclusion Criteria:

* age < 18 years or > 60 years
* diabetic history < 5 years
* BMI > 27
* body weight > 80 kg
* exogenous insulin requirement > 1 unit/kg/day
* severe anemia (male < 8 g/dl, female < 7 g/dl)
* low white blood cell count (< 3000/dl)
* liver dysfunction
* Active infection including hepatitis B, hepatitis C, HIV, or TB
* panel reactive antibody > 20%
* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Exogenous insulin requirement | 5
Hemoglobin A1c | 5
Glucose and C-peptide levels | 5

SECONDARY OUTCOMES:
liver function | 5
kidney function | 5
Portal vein Ultrasound | 1
autoantibodies | 5
Complete Blood Count | 5

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, professor, Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China